CLINICAL TRIAL: NCT00468442
Title: B-Lymphocyte Immunotherapy in Islet Transplantation: Toward Calcineurin-Inhibitor Free Immunosuppression (CIT-05)
Brief Title: B-Lymphocyte Immunotherapy in Islet Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CIT-05
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Insulin dependence; Hypoglycemia; Hypoglycemia unawareness
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Antilymphocyte Serum; Daclizumab; Rituximab; Sirolimus

ARMS (1):
- Allogeneic Pancreatic Islet Cells (Experimental): Participants will receive up to three islet transplants and maintenance immunosuppressive therapy.
  Interventions: Biological: Allogeneic Pancreatic Islet Cells; Biological: Antithymocyte globulin; Biological: Daclizumab; Biological: Rituximab; Drug: Sirolimus

INTERVENTIONS:
Biological: Allogeneic Pancreatic Islet Cells — transplant of islet cells injected into the portal vein of the liver
Biological: Antithymocyte globulin — Immunosuppressive that selectively depletes activated T-cells and depletes resting T-cells in a dose-dependent manner.
  Other Names: ATG
Biological: Daclizumab — Will replace antithymocyte globulin in all islet transplantations after the first one
  Other Names: Zenapax
Biological: Rituximab — Depletes transient B-cells
  Other Names: Rituxan
Drug: Sirolimus — Maintenance immunosuppressive therapy
  Other Names: Rapamune

SUMMARY:
Type 1 diabetes is an autoimmune disease in which the insulin-producing pancreatic beta cells are destroyed, resulting in poor blood sugar control. The purpose of this study is to determine the safety and effectiveness of islet transplantation, combined with the immunosuppressive medications and medications to support islet survival for treating type 1 diabetes in individuals experiencing hypoglycemia unawareness and severe hypoglycemic episodes.

DETAILED DESCRIPTION:
Type 1 diabetes is commonly treated with the administration of insulin, either by multiple insulin injections or by a continuous supply of insulin through a wearable pump. Insulin therapy allows long-term survival in individuals with type 1 diabetes; however, it does not guarantee constant normal blood sugar control. Because of this, long-term type 1 diabetic survivors often develop vascular complications, such as diabetic retinopathy, an eye disease that can cause poor vision and blindness, and diabetic nephropathy, a kidney disease that can lead to kidney failure. Some individuals with type 1 diabetes develop hypoglycemia unawareness, a life-threatening condition that is not easily treatable with medication and is characterized by reduced or absent warning signals for hypoglycemia. For such individuals, pancreas or pancreatic islet transplantation are possible treatment options. Unfortunately, insulin independence among islet transplant recipients tends to decline over time. New strategies aimed at promoting engraftment of transplanted islets are needed to improve the clinical outcomes associated with this procedure. The purpose of this study is to determine the safety and efficacy of islet transplantation, when combined with an immunosuppressive medication regimen containing rituximab. This regimen is intended to treat type 1 diabetes in individuals experiencing hypoglycemia unawareness and severe hypoglycemic episodes. This study will also seek to improve the understanding of determinants of success and failure of islet transplants for type 1 diabetes.

Eligible participants will be randomly assigned to this study or the Phase 3 islet transplantation study (DAIT CIT-07). Participants in this study will receive up to three separate islet transplants and a regimen of immunosuppressive medications consisting of antithymocyte globulin (ATG), sirolimus, and rituximab. They will begin receiving ATG, sirolimus, and rituximab 2 days prior to the first islet transplant. ATG will continue to be given until Day 2 post-transplant, and sirolimus will be given for the duration of the study. They will receive additional rituximab on Days 5 and 12 post-transplant.

Transplantations will involve an inpatient hospital stay and infusion of islets into the portal vein. Participants who do not achieve or maintain insulin independence by Day 75 post-transplant will be considered for a second islet transplant. Participants who remain dependent on insulin for longer than 1 month after the second transplant and who show partial graft function will be considered for a third islet transplant. Daclizumab or basiliximab will be used in place of ATG for the second and third transplants, if they are necessary. Participants who do not meet the criteria for a subsequent transplant and do not have a functioning graft will enter a reduced follow-up period.

There will be approximately 15 study visits following each transplant. A physical exam, review of adverse events, and blood collection will occur at most visits. A chest x-ray, abdominal ultrasound, electrocardiogram, quality of life questionnaires, urine collection, and glomerular filtrating rate (GFR) testing will occur at some visits. Participants will also test their own blood glucose levels at least four times per day throughout the study. A 12-month follow-up period will take place after the participant's last transplant.

ELIGIBILITY:
Inclusion Criteria:

* Mentally stable and able to comply with study procedures
* Clinical history compatible with type 1 diabetes with onset at less than 40 years of age, insulin dependence for at least 5 years at study entry, and a sum of age and insulin dependent diabetes duration of at least 28
* Absent stimulated C-peptide (less than 0.3 ng/ml) 60 and 90 minutes post-mixed-meal tolerance test
* Involvement of intensive diabetes management, defined as:

  1. Self-monitoring of glucose values no less than a mean of three times each day averaged over each week
  2. Administration of three or more insulin injections each day or insulin pump therapy
* Under the direction of an endocrinologist, diabetologist, or diabetes specialist with at least three evaluations the 12 months prior to study enrollment
* At least one episode of severe hypoglycemia in the past 12 months, defined as an event with one of the following symptoms: memory loss; confusion; uncontrollable behavior; irrational behavior; unusual difficulty in awakening; suspected seizure; seizure; loss of consciousness; or visual symptoms in which the participant was unable to treat him/herself and which was associated with either a blood glucose (BG) level < 54 mg/dL [3.0 mmol/L] or prompt recovery after oral carbohydrate, intravenous glucose, or glucagon administration, in the past 12 months prior to study enrollment
* Reduced awareness of hypoglycemia. More information about this criterion, including specific definition of hypoglycemia unawareness, is in the protocol.

Exclusion Criteria:

* Body mass index (BMI) greater than 30 kg/m2 or weight less than or equal to 50 kg
* Insulin requirement of more than 1.0 IU/kg/day or less than 15 U/day
* HbA1c greater than 10%
* Untreated proliferative diabetic retinopathy
* Systolic blood pressure higher than 160 mmHg or diastolic blood pressure higher than 100 mmHg
* Measured glomerular filtration rate using iohexol of less than 80 ml/min/1.73m2. More information about this criterion is in the protocol.
* Presence or history of macroalbuminuria (greater than 300 mg/g creatinine)
* Presence or history of panel-reactive anti-HLA antibody levels greater than 20% by flow cytometry. More information about this criterion is in the protocol.
* Pregnant, breastfeeding, or unwilling to use effective contraception throughout the study and 4 months after study completion
* Active infection, including hepatitis B, hepatitis C, HIV, or tuberculosis. More information about this criterion is in the protocol.
* Negative for Epstein-Barr virus by IgG determination
* Invasive aspergillus, histoplasmosis, or coccidioidomycosis infection within one year prior to study enrollment
* History of malignancy except for completely resected squamous or basal cell carcinoma of the skin
* Known active alcohol or substance abuse
* Baseline Hgb below the lower limits of normal, lymphopenia, neutropenia, or thrombocytopenia
* History of Factor V deficiency
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy after transplantation or individuals with an INR greater than 1.5
* Severe coexisting cardiac disease, characterized by any one of the following conditions:

  1. Heart attack within the last 6 months
  2. Evidence of ischemia on functional heart exam within the year prior to study entry
  3. Left ventricular ejection fraction less than 30%
* Persistent elevation of liver function tests at the time of study entry
* Symptomatic cholecystolithiasis
* Acute or chronic pancreatitis
* Symptomatic peptic ulcer disease
* Severe unremitting diarrhea, vomiting, or other gastrointestinal disorders that could interfere with the ability to absorb oral medications
* Hyperlipidemia despite medical therapy (fasting LDL cholesterol greater than 130 mg/dl, treated or untreated; and/or fasting triglycerides greater than 200 mg/dl)
* Receiving treatment for a medical condition that requires chronic use of systemic steroids, except the use of 5 mg or less of prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only
* Treatment with antidiabetic medication other than insulin within the past 4 weeks
* Use of any investigational agents within the past 4 weeks
* Received a live attenuated vaccine(s) within 2 months of study entry
* Any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial
* Treatment with any immunosuppressive regimen at the time of enrollment
* A previous islet transplant
* A previous pancreas transplant, unless the graft failed within the first week due to thrombosis, followed by pancreatectomy and transplant occurred more than 6 months prior to enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Insulin independence | 75 days after a single islet transplant

SECONDARY OUTCOMES:
reduction in insulin requirements, HbA1c, MAGE, LI, HYPO score, fasting glucose, beta score, quality of life | 75 days and 1 year following first and final infusion

CONTACTS AND LOCATIONS:
Overall Officials: Ali Naji, MD, PhD, Study Chair — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Click here for the Clinical Islet Transplantation Consortium Web site — http://www.citisletstudy.org
- See also: Click here for more information about the University of Pennsylvania's Type 1 Diabetes Unit — http://www.med.upenn.edu/idom/t1diabetes.html